CLINICAL TRIAL: NCT05840575
Title: A Multidisciplinary Neuroscience Approach to Investigate Cognitive Impairment in Young Patients With Cancer Prospectively
Brief Title: Investigating Cognitive Impairment in Young Patients With Cancer Prospectively
Acronym: MyBrain
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lisa Lyngsie Hjalgrim, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: MyBrain
Record Dates: First submitted 2023-01-25; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Chemotherapy-Related Cognitive Impairment; Chemotherapeutic Toxicity; Chemo-brain; Cancer; Childhood Cancer; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Testicular Cancer; Sarcoma; Leukemia
Keywords: Cognition; Neuropsychology; Electroencephalogram; Biomarkers
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Testicular Neoplasms; Sarcoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Solid tumor patients: Patients diagnosed with solid tumor cancers
- Haematological patients: Patients diagnosed with haematological cancers

SUMMARY:
The MyBrain study investigates the brain function of children, adolescents and young adults during and after chemo treatment for cancer. The tests include 1) cognitive skills such as memory and attention; 2) the brain's electrical activity; 3) and biological markers related to brain function.

The aim of the study is to better understand the trajectories of cognitive functioning and measures that have been associated with cognitive impairment in patients treated with chemotherapy.

DETAILED DESCRIPTION:
Background:

Numerous studies indicate that many patients with cancer, regardless of cancer type, develop cancer-related cognitive impairment (CRCI), which may persist for many years after ended treatment. CRCI can occur regardless of cancer type and most often affects cognitive domains, such as memory, attention processing speed, and executive functions. In daily life, this may manifest as difficulties in attention and concentration, learning, multitasking, mentally organize tasks, and cognitive fatigue. The cognitive impact of cancer and cancer treatments for non-CNS patients has been shown with several research disciplines, such as neuropsychological tests, neuroimaging, biomarkers, and animal studies.

Cognitive impairment affects children, adolescents, and young adults with cancer and their families. Young cancer patients may be particularly vulnerable to cognitive impairment as the brain undergoes development in childhood and continues into the twenties. However, there is a lack of knowledge about when a decrease in cognitive capacity may occur, how long it will persist, and which cognitive domains are affected for children adolescents and young adults with cancer.

Aim:

MyBrain is an explorative study which will explore and describe trajectories of CRCI as measured by neuropsychological assessment, self-reported quality of life and fatigue, brain functioning measured with electroencephalogram (EEG), and biomarkers of neural impairment and inflammation.

Design:

Single-centre, prospective longitudinal study including patients diagnosed with cancers outside the brain at age 7-29 years. Each patient is paired with a healthy control matched on age and social circle.

Time points:

The MyBrain study includes patients with different cancer types and assigned to different treatment protocols. Therefore, some patients will undergo treatment for several months (for instance testicular cancer, lymphomas), while others will be treated over several years (acute lymphoblastic leukaemia). The measurement time points will vary between different protocols.

T0: Patients are assessed as close to the day of diagnosis as possible, within 30 days from the day they receive their diagnosis.

T1abc: Up to three time points (2-3) during chemo treatment. Blood samples will be taken immediately before and 10-14 days after the chemo dosing for the specific chemo cycles. For patients who receive more than three cycles of chemotherapy, the timepoints T1abc, will be placed at the chemo treatments with the highest doses (denoted the major chemo treatments) according to the treatment protocol the patient follows. If the treatment protocol allocates the same dose to all chemo treatments, the T1abc will be placed with the aim to obtain approximate equidistance between T0, T1abc and T2.

HDM1-3: Three additional time points during treatment for the patients who are treated with high dose methotrexate (HDM). Blood samples will be taken immediately before and 10-14 days after HDM treatment.

T2: End of treatment. End of treatment is defined as two weeks after the final antineoplastic treatment. For ALL patients, end of treatment is defined as the end of consolidation treatment.

T3: Follow-up, 6 months after T2.

All outcome measures are collected at the time points T0, T2 and T3 for patients and at similar time intervals for controls. T1abc and HDM1-3 only includes biological samples from the patients.

Data includes:

* Clinical information obtained from medical charts including cancer diagnosis, treatment protocol, duration of treatment and adverse events.
* Sociodemographic information collected with a brief questionnaire which includes level of education, occupation, economic status, and the parents' level of education and occupation.
* Cognitive functioning assessed with a clinical battery. The battery includes: Nepsy-II Verbal Fluency, Wechsler Coding (WISC-V or WAIS-IV), Wechsler Symbol Search (WISC-V or WAIS-IV), RBANS Word List Memory, RBANS Word List memory recall, RBANS Word List memory recognition, Wechsler Vocabulary (WISC-V or WAIS-IV), Wechsler Matrix (WISC-V or WAIS-IV), Digit Span (WISC-V or WAIS-IV), Conner´s CPT-III, Grooved Pegboard. For the Wechler tests, participants <16 years of age are tested with WISC-V and participants 16 or older are tested with WAIS-IV.
* Cognitive functioning assessed with the Cambridge Neuropsychological Test Automated Battery (CANTAB). The following tests are included: Spatial Working Memory, Pattern Recognition Memory, Spatial Span, Paired Associates Learning, Pattern Recognition Memory (delayed), Delayed Matching to Sample.
* Qualitive of life measured with the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scales 4.0
* Fatigue measured with the PedsQL Multidimensional Fatigue Scales 3.0
* Resting state EEG is recorded with eyes-open (EO) and eyes-closed (EC) in four blocks of three minutes each (EO-EC-EO-EC).
* Event-related potentials (ERP) during a two-tone auditory oddball task. The participants are instructed to mentally count the rare stimulus.
* Biomarkers of associated with cognitive functioning, measured in serum: neurofilament light chain, glial fibrillary acidic protein, brain derived neurotrophic factor, and pro- and anti-inflammatory markers (IFNy, IL10, IL12p70, IL17A, IL6, TNFa and IL1β).
* Biomarkers of associated with cognitive functioning, measured in cerebrospinal fluid (CSF) for the haematological patients if CSF is drawn as part of their treatment: neurofilament light chain, glial fibrillary acidic protein, brain derived neurotrophic factor, pro- and anti-inflammatory markers.

Data analyses Large inhomogeneity in the data is expected due to the inclusion of patients over a wide age-span with different cancer types, varying treatment protocols, and varying timelines from diagnosis to end of treatment and there are no predefined, specific hypotheses due to the many sources of inhomogeneity. All analyses are exploratory, and confidence limits (rather than nominal p-values) will be used as the indication of the strength of an association when quantified in statistical analyses.

The initial analyses will be data visualizations of quantitative variables will include trajectories for single variables, bivariate plots with smoothed mean curves added, and plots of patient observations against the corresponding observations for the matched control connecting the points in temporal order for each matched pair. The trajectories will be presented for different timescales, e.g., time since diagnosis, or time from T2. Potential risk factors, like cancer type, sex, or age will be indicated in the data visualizations by using different colours and symbols.

Neurocognitive test scores will be investigated at each time point (T0, T2, and T3) for each subtest. Raw as well as scaled scores, age-adjusted from Danish population norms, will be used in the analysis. For the visualizations of the raw test scores, the scores will be plotted as a function of age including reference curves based on back-converted means, ±SD, and -2 SD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly diagnosed with a non-CNS cancer and will undergo chemotherapy at University Hospital Copenhagen, Rigshospitalet.
* At the age of 7-29 years at diagnosis
* Each patient is matched (1:1) with a control participant within 24 months of age. The controls are recruited from the patient's own social circle and can be a friend, partner, or close family (sibling or cousin).

Exclusion Criteria:

* Unable to speak and understand Danish
* Severe intellectual disability or mental health disorder that hinders participation
* Brain metastases,
* Terminal illness
* Have had a previous chemotherapy or radiotherapy treatment

Ages: 7 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who are diagnosed with a non-central nervous system cancer at Rigshospitalet in Copenhagen, Denmark. The distribution of different cancer diagnoses in the study population will reflect the distribution of non-CNS diagnoses among patients in the age group receiving chemotherapy at the study site. The most common diagnoses are Hodgkin lymphoma, non-Hodgkin lymphoma, testicular cancer, sarcoma, and leukaemia. Approximately 30-40 new patients are expected to be included every year (in total 100 patients during the three-year recruitment period).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Performance on clinical neurocognitive tests: Wechlers scale | T0: within 30 days of diagnosis
  Scores on the clinical neurocognitive tests (Wechler Intelligence Scale for Children Fifth edition for participants 7-15.9 years of age, Wechler Adult Intelligence Scale Fourth edition for participants 16 years of age or older). Scaled scores range from 0-19, higher = better performance.
Performance on clinical neurocognitive tests: Wechlers scale | T2: end of treatment (2 weeks after the final antineoplastic treatment)
  Scores on the clinical neurocognitive tests (Wechler Intelligence Scale for Children Fifth edition for participants 7-15.9 years of age, Wechler Adult Intelligence Scale Fourth edition for participants 16 years of age or older). Scaled scores range from 0-19, higher = better performance.
Performance on clinical neurocognitive tests: Wechlers scale | T3: 6 months after end of treatment
  Scores on the clinical neurocognitive tests (Wechler Intelligence Scale for Children Fifth edition for participants 7-15.9 years of age, Wechler Adult Intelligence Scale Fourth edition for participants 16 years of age or older). Scaled scores range from 0-19, higher = better performance.

SECONDARY OUTCOMES:
Trajectories of performance on clinical neurocognitive tests: Grooved Pegboard test | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  The Grooved Pegboard (Lafayette Instrument) is a neurocognitive test consisting of consisting of key shapes (pegs) and matching holes used to test visual-motor coordination. Scores are in milliseconds, lower scores = better performance.
Trajectories of performance on clinical neurocognitive tests: Repeatable Battery for the Assessment of Neuropsychological Status | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) subtests List Learning, List Recall and List Recognition evaluates learning and memory. Scaled scores (t-scores) range from 0-100, higher = better performance.
Trajectories of performance on clinical neurocognitive tests: Conner's Continuous Performance Test | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  The Conner's Continuous Performance Test Third edition evaluates attention-related performance in areas of inattentiveness, impulsivity, sustained attention, and vigilance. Scaled scores (t-scores) range from 0-100, higher = better performance.
Trajectories of performance on clinical neurocognitive tests: NEPSY-II, A Developmental Neuropsychological Assesment of Neuropsychological Status | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  The NEPSY Second edition Verbal Fluency subtest is used to evaluate executive and verbal cognitive skills. The scores are the number of correct words generated for the two semantic and two lexical fluency tasks, rang 0-no upper limit, more words = higher score.
Trajectories of performance on automated cognitive tests | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Neuropsychological functions measured with the Cambridge Neuropsychological Test Automated Batteries(CANTAB), using the subtests Spatial Working Memory, Pattern Recognition Memory, Spatial Span, Paired Associates Learning, Pattern Recognition Memory (delayed), Delayed Matching to Sample. The tests can generate several outcomes, % of correct responses will primarily be used (0-100, higher = better performance).
Trajectories of quality of life | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Pediatric Quality of Life Inventory Generic Core Scales 4.0 (5-point Likert scale from 0 (Never) to 4 (Almost always), lower meaning better outcome).
Trajectories of fatigue | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Pediatric Quality of Life Inventory Multidimensional Fatigue Scales 3.0 (5-point Likert scale from 0 (Never) to 4 (Almost always), lower meaning better outcome).
Trajectories of resting-state EEG: the power spectrum, absolute delta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Absolute power (microvolts squared) in the delta band.
Trajectories of resting-state EEG: the power spectrum, absolute theta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Absolute power (microvolts squared) in the theta band.
Trajectories of resting-state EEG: the power spectrum, absolute alpha power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Absolute power (microvolts squared) in the alpha band.
Trajectories of resting-state EEG: the power spectrum, absolute beta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Absolute power (microvolts squared) in the beta band.
Trajectories of resting-state EEG: the power spectrum, relative delta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Relative power (%) in the delta band.
Trajectories of resting-state EEG: the power spectrum, relative theta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Relative power (%) in the theta band.
Trajectories of resting-state EEG: the power spectrum, relative alpha power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Relative power (%) in the alpha band.
Trajectories of resting-state EEG: the power spectrum, relative beta power | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Relative power (%) in the beta band.
Trajectories of the ERP oddball test: P300 amplitude | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Amplitude (in microvolts) of the P300 peak.
Trajectories of the ERP oddball test: P300 peak latency | T0: within 30 days of diagnosis, T2: end of treatment (2 weeks after the final antineoplastic treatment); T3: 6 months after end of treatment
  Latency (in microseconds) of the P300 peak.
Trajectories of serum levels of biomarkers of neurodegeneration and inflammation | T0: within 30 days of diagnosis; T1acb: immediately before and 10-14 days after major chemo treatments, HDM1-3 immediately before and 10-14 days after HDM; T2: end of treatment (2 weeks after final antineoplastic treat.); T3: 6 months after end of treat.
  Concentration (pg/ml) of neurofilament light chain, glial fibrillary acidic protein, brain derived neurotrophic factor, pro- and anti-inflammatory markers (IFNy, IL10, IL12p70, IL17A, IL6, TNFa and IL1β).
Trajectories of cerebrospinal fluid levels of biomarkers of neurodegeneration and inflammation | T0: within 30 days of diagnosis; T1acb: immediately before and 10-14 days after major chemo treatments, HDM1-3 immediately before and 10-14 days after HDM; T2: end of treatment (2 weeks after final antineoplastic treat.); T3: 6 months after end of treat.
  Concentration (pg/ml) of neurofilament light chain, glial fibrillary acidic protein, brain derived neurotrophic factor, pro- and anti-inflammatory markers (IFNy, IL10, IL12p70, IL17A, IL6, TNFa and IL1β).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordhjem BJT, Tjornlund M, Thomsen BL, Hjerming M, Kjaer TW, Pappot H, Hjalgrim LL. Protocol for a prospective, longitudinal study of cognitive impairment in young patients with cancer: a multidisciplinary neuroscience approach (MyBrain). BMJ Open. 2023 May 18;13(5):e070534. doi: 10.1136/bmjopen-2022-070534. PMID 37202143
- See also: Project website — https://mybrain.nu
- See also: Department website — https://www.rigshospitalet.dk/english/departments/juliane-marie-centre/